CLINICAL TRIAL: NCT00003359
Title: Phase I Dose Escalation Study to Evaluate the Safety of T138067-Sodium in Patients With Advanced Refractory Cancer
Brief Title: T138067 Sodium in Treating Patients With Advanced Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-004; CDR0000066341 (Registry Identifier: PDQ (Physician Data Query)); TULA-T9801; NCI-G98-1443
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Drug: batabulin sodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of T138067 sodium in treating patients with advanced refractory cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of T138067 sodium that can be given to patients with advanced refractory cancer on a 28-day schedule and establish a dose for further study. II. Evaluate the safety and dose limiting toxicity of T138067 sodium in these patients. III. Determine the pharmacokinetic parameters after a single intravenous dose of this agent in these patients. IV. Obtain safety data and preliminary efficacy information after repetition of single doses of T138067 sodium in these patients.

OUTLINE: This is an open label, dose escalation study. Patients receive T138067 sodium by IV over 3 hours. Patients may be retreated every 4 weeks for up to 6 courses (6 months total) in the absence of disease progression or dose limiting toxicity (DLT). At least 3 patients are treated at each dose level in the absence of DLT. The maximum tolerated dose is defined as the dose level where 2 of 3-6 patients experience DLT.

PROJECTED ACCRUAL: Approximately 3-24 patients will be accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced refractory cancer Must meet one of the following criteria: - Failed at least 1 regimen of radiotherapy, chemotherapy, or immunotherapy and not a candidate for a regimen of higher efficacy - Refractory to existing standard therapy and not candidate for a regimen of higher efficacy - Advanced malignancy for which there is no standard chemotherapy available No known brain metastases or leptomeningeal involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Greater than 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Prothrombin time at least 30% of control Partial thromboplastin time at least 30% of control Hepatic: Bilirubin less than 2 mg/dL ALT and AST no greater than 2 times normal Alkaline phosphatase no greater than 2 times normal Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No New York Heart Association class III or IV heart disease No myocardial infarction in the past 6 months Other: No immunodeficiency syndrome (acquired or congenital) No uncontrolled infection No significant comorbidity that may compromise participation in this study Not pregnant Effective contraception required of all fertile patients during and until 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 4 weeks since prior immunotherapy No concurrent immunotherapy or biologic response modifier therapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy No concurrent chemotherapy Endocrine therapy: No concurrent corticosteroids Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: At least 3 weeks since any prior major surgery Other: No organ allograft At least 30 days since any prior investigational agents No concurrent nonsteroidal antiinflammatory agents or aspirin No concurrent alternative therapies (i.e., herbal medicines, high doses of vitamins) No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1998-04; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spriggs, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Background] Jahan TM, Sandler A, Burris H, et al.: A phase II study of T138067-sodium in prior taxane-treated patients (pts) with locally advanced or metastatic non-small cell lung cancer (NSCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1282, 2002.